CLINICAL TRIAL: NCT03296982
Title: A Study to Determine the Inter/Intra Observer and Intra-Subject Variability of Whole Blood Clotting Time Measurements in Ex Vivo Human Blood Samples Spiked With Anticoagulants
Brief Title: Variability of Whole Blood Clotting Time Measurements in Ex Vivo Human Blood Samples Spiked With Anticoagulants
Status: Completed | Type: Observational
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Other Study IDs: PER977-01-010
Record Dates: First submitted 2014-12-18; First posted 2017-09-29 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Whole blood clotting time
MeSH Terms: interventions — edoxaban; Enoxaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood Sample: Blood will be sampled by direct venipuncture on 8 occasions.
  Interventions: Other: Blood drawn by direct venipuncture; Drug: edoxaban; Drug: Enoxaparin; Drug: Saline sham

INTERVENTIONS:
Other: Blood drawn by direct venipuncture — Subjects will have blood sampled (12 mL/sample) a total of 8 times by direct venipuncture. Samples will be spiked with predetermined concentrations of anticoagulants, or saline sham.
Drug: edoxaban
Drug: Enoxaparin
Drug: Saline sham

SUMMARY:
The study will assess the distribution and variability of whole blood clotting time (WBCT) measurement in human blood collected from healthy volunteers that is untreated and spiked with predetermined concentrations of edoxaban or enoxaparin.

DETAILED DESCRIPTION:
Twelve healthy volunteers aged 18 to 65 years (6 subjects per spiking anticoagulant) will be enrolled. A total of 8 blood samples (12 mL/sample) will be collected by direct venipuncture. The samples from will be spiked with predetermined concentrations of edoxaban or enoxaparin (baseline, saline control and 6 specified concentrations of anticoagulant).

Each blood sample will be tested for whole blood clotting time (WBCT), Point of Care activated partial thromboplastin time (aPTT) and prothrombin time (PT).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form
2. Healthy male and female subjects aged 18 to 65 years (inclusive) with suitable veins for venipuncture -

Exclusion Criteria:

1. Subjects who cannot communicate reliably with the Investigator
2. History of major bleeding or major trauma within the 6 months prior to signing informed consent
3. Propensity to bleeding (i.e. due to recent trauma, surgery, peptic ulcer, gastrointestinal bleeding or hemorrhoids)
4. Significant infection or known inflammatory process in the 2 weeks prior to screening
5. Active smoker or current use of any tobacco products or use within 3 months prior to signing informed consent
6. Treatment with any investigation product or therapy within 30 days prior to screening
7. Received non-steroidal antiinflammatory drugs or medications (including anticoagulants or aspirin) with a direct effect on hemostasis within 7 days of blood sampling
8. Unwilling to comply with the procedures in the protocol
9. Currently enrolled in any other study -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Distribution and variability of WBCT measurements | 1 day
  Assessment of the analytical measurement range, reproducibility and precision of WBCT measurement in human blood spiked with predetermined concentrations of enoxparin and edoxaban

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Quintiles Phase 1 Services, LLC Overland Park KS